CLINICAL TRIAL: NCT03701360
Title: Anti-platelet Precision Medicine to Prevent Stroke Early Progression and Recurrence (PRECISE)
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dong-Wha Kang, Principal Investigator, Asan Medical Center
Other Study IDs: PRECISE
Record Dates: First submitted 2018-09-14; First posted 2018-10-10 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspirin alone group: - Aspirin: 75~100mg once per day, initial loading dose of 300~500mg/d is allowed
- Aspirin + Clopidogrel resinate group: * Aspirin: 75~100mg once per day, initial loading dose of 300~500mg/d is allowed
  * Clopidogrel resinate: 75mg once per day, initial loading dose of 300mg/d is allowed

SUMMARY:
This is a pragmatic, multi-center, non-interventional, non-randomized prospective observational study.

DETAILED DESCRIPTION:
This is a prospective study of patients with acute stroke or transient ischemic attack within 72 hours of symptom onset. It is to mainly observe the patients' prognosis following the prescription of clopidogrel resinate and aspirin, collect relevant data and create big data for stroke. Based on this data, an AI, using various advanced statistical methodologies and deep learning techniques will be developed, and offer information regarding stroke prognosis by extracting markers that are characteristic of the relationship between stroke and the study drug.

These analyses and results will include information on which drug regimen will better prevent the progression or recurrence of stroke by considering individual patient conditions. This is a pragmatic trial based on the prescription and treatment processes of routine clinical practice. Thus, there is no major restriction and with only the minimum exclusion criteria in place, it does not hinder usual clinical practices. Therefore, selecting and changing a patient's antiplatelet agents should be a rational medical judgment made by the patient's attending physician. The study will proceed without any major change in the sequence of routine clinical examinations, prescriptions, treatments, observations, etc. Provided, the process of storing and analyzing relevant information will be added to each study procedure in accordance with study methodologies and conditions no other special efforts or limitations will be required.

The data will be collected prospectively, and the AI will generate brain imaging data and prognostic indicators for 3-months after stroke has occurred. The performance of the AI will be verified with independent test sets.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects who are aged 19 or over.
2. Patients with acute non-cardiac stroke or transient ischemic attack within 72 hours of the onset (in the case of a transient ischemic attack, presence of ischemic/ischemic lesion on DWI or PWI).
3. Patients whose informed consent document within 72 hours of onset was signed and submitted.
4. Patients who were treated with aspirin alone or aspirin plus clopidogrel resinate following stroke.

Exclusion Criteria:

1. Patients who need anticoagulants for cardiac ischemic stroke or other reasons.
2. Patients who suffered severe stroke (National Institutes of Health Stroke Scale> 16).
3. Patients who received emergency remission therapies such as tPA and thrombolysis.
4. Patients with neurological deterioration prior to signing an informed written consent document.
5. Patients who have undergone patency procedures (surgery or stent insertion) in the cerebrovascular or carotid arteries following stroke or are expected to do so.
6. Patients who are scheduled to undergo major surgery.
7. Patients who developed stroke during procedure/surgery.
8. Patients with recent history (in the past three months) of cerebral hemorrhage.
9. Patients with active internal bleeding.
10. Patients with severe anemia (Hb <10 g / dL) or bleeding tendency (platelet <100,000 / uL or PT-INR> 1.7).
11. When a patient's life expectancy is less than 6 months due to other systemic disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients:
  Transient ischemic attack with confirmed acute ischemic stroke by brain imaging
Sampling Method: Probability Sample
Enrollment: 1199 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Rate of patients with neurological deterioration under hospital treatment. | up to 3 months after stroke onset
  Rapid worsening of an existing focal neurological deficit or rapid onset of a new focal neurological deficit (≥ 24 hours) that is clinically judged by the Investigator not to be attributable to non-ischemic etiology.
Rate of patients with new ischemic stroke under hospital treatment. | up to 3 months after stroke onset
  * Rapid onset of a new focal neurological deficit with clinical or imaging evidence of infarction and not attributable to a non-ischemic etiology (not associated with brain infection, trauma, tumor, seizure, severe metabolic disease, or degenerative neurological disease); or,
  * Rapid worsening of an existing focal neurological deficit that is judged by the Investigator to be attributable to a new infarction. Criteria for symptoms attributable to new infarction may include symptoms that persist and are judged by the investigator to be attributable to new infarction, imaging evidence of infarction, or no evidence of a non-ischemic etiology.
Rate of patients with symptomatic hemorrhagic transformation of an ischemic stroke under hospital treatment. | up to 3 months after stroke onset
  Imaging evidence (by CT or MR) of extravascular blood within the area of infarction, and symptoms judged to be related to the hemorrhagic transformation.
  Scenarios which may be judged as symptomatic:
  * If blood is already present on imaging at presentation, symptoms are out of proportion to what would be expected for the size and location of the infarct at presentation;
  * Clinical deterioration, defined by an increase of 4 points or more in the score on the NIHSS or leading to death, occurring after the initial ischemic event, and identified as the result of the hemorrhagic transformation; or
  * Mass effect secondary to the hemorrhagic transformation causing symptoms.
Rate of patients with symptomatic intracranial hemorrhage under hospital treatment. | up to 3 months after stroke onset
  Evidence of hemorrhage in the brain parenchyma or extraparenchymal spaces demonstrated by head imaging, surgery, or autopsy, which is not in the same territory of an underlying acute or subacute ischemic stroke, and is judged to be associated with any new neurologic symptoms (including headache) or leading to death.
Rate of patients with myocardial infarction under hospital treatment. | up to 3 months after stroke onset
  The diagnosis of MI will be based on an algorithm developed from the Universal Definition of Myocardial Infarction (Circulation 2007 116:2634-2653) that takes into account 5 categories of clinical information from the acute event: rise and/or fall of cardiac biomarkers, ECG abnormalities, clinical setting, imaging evidence, and pathology.
Rate of patients with coronary revascularization without myocardial infarction under hospital treatment. | up to 3 months after stroke onset
  Documented coronary angioplasty, stenting, or bypass surgery for demonstrated or presumed coronary artery disease.
Rate of patients with major hemorrhage other than intracranial hemorrhage under hospital treatment. | up to 3 months after stroke onset
  A hemorrhagic event, judged to be nontraumatic, that results in intraocular bleeding causing loss of vision, the need for a transfusion of two or more units of red cells or the equivalent amount of whole blood, or the need for hospitalization or prolongation of existing hospitalization. This may include bleeding events related to surgical procedures but not those related to accidental trauma. Life-threatening hemorrhagic events will be defined as those that are fatal or require use of intravenous inotropic medication to maintain blood pressure, interventional treatment (including surgical, endoscopic or endovascular interventions), or transfusion of four or more units of red cells or the equivalent amount of whole blood. Non-life-threatening hemorrhagic events will be defined as those classified as major hemorrhagic events but not as life-threatening.
Rate of patients with minor hemorrhage other than intracranial hemorrhage under hospital treatment. | up to 3 months after stroke onset
  All hemorrhagic events leading to interruption of therapy or discontinuation of the study drug but not classifiable as major hemorrhagic events. This may include bleeding events related to surgical procedures but not those related to accidental trauma.
Rate of patients with ischemic vascular death under hospital treatment. | up to 3 months after stroke onset
  Death due to ischemic stroke, myocardial infarction, sudden cardiac death, arrhythmia, pulmonary embolism, bowel or limb infarction, or any death not readily attributable to a non-ischemic cause.
Rate of patients with hemorrhagic vascular death under hospital treatment. | up to 3 months after stroke onset
  Death due to intracranial or systemic hemorrhage.
Rate of patients with other serious adverse event under hospital treatment. | up to 3 months after stroke onset
  Any adverse event, not belonging to the other outcome event categories, that is fatal or life threatening, is permanently or substantially disabling, requires or prolongs hospitalization, results in a congenital anomaly, or requires intervention to prevent permanent impairment or damage.

SECONDARY OUTCOMES:
Evaluation by an independent investigator | up to 3 months after stroke onset
  A direct comparison between the aspirin alone group and the aspirin plus clopidogrel group for the incidence of 11 outcome variables evaluated by an independent investigator at the primary endpoints will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wha Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Dong-Wha Kang, Seoul, South Korea

DOCUMENTS (1):
  • Study Protocol (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03701360/Prot_000.pdf